CLINICAL TRIAL: NCT04631432
Title: Choice Switching and Autism
Status: Completed | Type: Observational
Sponsor: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Eldad Yechiam, Professor, Technion, Israel Institute of Technology
Other Study IDs: 109171; Technion institute 109171 (Other Grant/Funding Number: Technion - Israel Institute of Technology)
Record Dates: First submitted 2020-11-04; First posted 2020-11-17 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Autism Spectrum Disorder; Decision Making
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participation: All participants will complete the same protocol
  Interventions: Diagnostic Test: Pre-screening; Behavioral: Task session

INTERVENTIONS:
Diagnostic Test: Pre-screening — Document upload of Autism diagnosis certificate. Participants can request to show their certificate via a Zoom meeting with the researcher instead of uploading it.
Behavioral: Task session — The Iowa Gambling task- four decks of cards on the computer screen. Each card yields a reward, but might also yield a loss. In each trial, the participant selects a card. Consequently, the card is exposed, displaying the gain and the loss for that trial. Through contingent feedback, participants are expected to learn that some deck are better than others.The task will include 120 trials.
  Block of trials without feedback- four decks of cards on the computer screen. Each card yields a reward, but might also yield a loss. In each trial, the participant selects a card. Consequently, the card is exposed, but the gain and the loss for that trial are not displayed. The task will include 30 trials.
  Social Responsiveness Scale, 2nd Edition (SRS-2; adult-self report):(Constantino & Gruber, 2012) The brief autism quotient scale:(AQ10; Baron-Cohen et al., 2001) Brief intelligence test (Similarities-MAB + Raven Set 1)

SUMMARY:
The study aims to replicate and clarify a recently observed phenomenon whereby individuals with Autism Spectrum Disorder (ASD) switch between options in a repeated task to a greater extent than healthy controls do. In a meta-analysis a large effect size was found (.37) yet because the effect was noisy in different studies it was not statistically significant. The investigators seek to first examine a very large population through an Internet mediated platform. The sample size will be about the size of all of the previous studies that examined this issue together. Secondly, the investigators wish to understand the discrepancy between this choice switching phenomenon and the recorded tendency of ASD individuals to avoid changing choices. First, the investigators will administer the task in which the effect was found (the Iowa Gambling task) for a longer duration than previously and evaluate whether ASD individuals show increased choice switching in the first blocks of trials but reduced switching following more experience. Secondly, the investigators will administer an additional block of trials without feedback in which participants will not be able to go through a learning process. The investigators predict that this will reduce (and possible flip) the tendency of individuals with ASD to switch choices more often.

ELIGIBILITY:
Inclusion Criteria:

* ASD group - Diagnosed with ASD
* Control - No ASD diagnosis: within age and education range of the ASD group.

Exclusion Criteria:

* Demographics: Under 18 years of age.
* Mental health: self reported brain injury and neurological disorder (besides autism).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Same proportion of males and females from the two groups.
Study Population: We will recruit participants using websites for recruiting experimental participants worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Mean run size | Through study completion, an average of 1 year
  Number of consecutive selections from the same deck (across trials and in different blocks).
Advantageous selections | Through study completion, an average of 1 year
  Percentage of advantageous selections(across trials and in different blocks).

CONTACTS AND LOCATIONS:
Overall Officials: Dana Zeif, MSc, Study Director — Technion, Israel Institute of Technology; Ofir Yakobi, PhD, Study Director — University of Waterloo; Eldad Yechaim, Professor, Principal Investigator — Technion, Israel Institute of Technology
Locations (1):
- Technion, Israel Institute of Technology, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeif D, Yechiam E. Autism is not associated with poor or enhanced performance on the Iowa Gambling Task: A Meta-Analysis. Neurosci Biobehav Rev. 2020 Jun;113:440-447. doi: 10.1016/j.neubiorev.2020.04.016. Epub 2020 Apr 18. PMID 32311370
- [Background] Bechara A, Damasio AR, Damasio H, Anderson SW. Insensitivity to future consequences following damage to human prefrontal cortex. Cognition. 1994 Apr-Jun;50(1-3):7-15. doi: 10.1016/0010-0277(94)90018-3. PMID 8039375
- [Background] Ozonoff S. Reliability and validity of the Wisconsin card sorting test in studies of autism. Neuropsychology. 1995;9(4):491.
- [Background] Gaeth GJ, Levin IP, Jain G, Data EV. Toward understanding everyday decision making by adults across the autism spectrum. Judgment and Decision Making. 2016 Nov 1;11(6):537.
- Available data/document: Statistical Analysis Plan — https://docs.google.com/document/d/16IlMPOgJMoh8tLIhB4JK5yeHI-0MfJVvRnQ8PdNp8-o/edit?usp=sharing
- Available data/document: Study Protocol — https://drive.google.com/file/d/1YoXgB4ifoeu2Z8OnG6_hVWP4sBLRp9wP/view?usp=sharing
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1WHJz01_y_b-gO4ZpZNAQsnqNf_SwdwNX/view?usp=sharing